CLINICAL TRIAL: NCT07150208
Title: Trastuzumab Deruxtecan With or Without Bevacizumab for HER2-low Unresectable and/or Metastatic Breast Cancer With Brain Metastasis: A Multicenter, Randomized, Open Label, Phase II Trial (THUMB Trial)
Brief Title: T-DXd With or Without Bevacizumab for HER2-low Breast Cancer With Brain Metastasis
Acronym: THUMB
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC- N0102
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer With Brain Metastasis; HER2-low Expressing Breast Cancer
Keywords: Breast Cancer with Brain Metastasis; HER2-low Expressing Breast Cancer; Trastuzumab Deruxtecan; Bevacizumab
MeSH Terms: interventions — Bevacizumab; trastuzumab deruxtecan

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T-DXd (Active Comparator): T-DXd: 5.4mg/kg intravenously (IV) every 3 weeks (Q3W).
  Interventions: Drug: Trastuzumab Deruxtecan (T-DXd)
- T-DXd+Bevacizumab (Experimental): T-DXd: 5.4mg/kg intravenously (IV) every 3 weeks (Q3W). Bevacizumab: 15mg/kg intravenously (IV) every 3 weeks (Q3W).
  Interventions: Drug: Bevacizumab (Bev); Drug: Trastuzumab Deruxtecan (T-DXd)

INTERVENTIONS:
Drug: Bevacizumab (Bev) — Bevacizumab is a drug that targets vascular endothelial growth factor (VEGF) and inhibits tumor angiogenesis, thereby inhibiting tumor growth and spread. In the treatment of breast cancer, Bevacizumab can be used in combination with chemotherapy to improve treatment outcomes and extend patients' progression-free survival and overall survival.
  Other Names: HLX04
  Arms: T-DXd+Bevacizumab
Drug: Trastuzumab Deruxtecan (T-DXd) — Trastuzumab deruxtecan (T-DXd) is an antibody-drug conjugate (ADC) composed of an anti-HER2 monoclonal antibody (trastuzumab), a cleavable linker, and a topoisomerase I inhibitor (an exatecan derivative). It targets and binds to HER2-positive tumor cells, internalizes, and releases cytotoxic drugs to induce DNA damage and apoptosis. It also has a "bystander effect" that can kill neighboring tumor cells with low HER2 expression, enhancing anti-tumor activity. T-DXd has shown significant efficacy in HER2-positive advanced breast cancer, with key clinical trials (such as DESTINY-Breast03) confirming that its progression-free survival (PFS) and overall survival (OS) are superior to traditional second-line treatments, with a median PFS reaching 28.8 months. Additionally, for HER2-low-expressing (IHC 1+ or 2+/ISH-) metastatic breast cancer (in the DESTINY-Breast04 study), T-DXd can extend PFS and OS, becoming the first targeted therapy to alter the survival outcomes of such patients.
  Other Names: DS8201

SUMMARY:
A phase II, open-label, multicenter, randomized controlled trial exploring the efficacy and safety of Trastuzumab Deruxtecan combined with or without Bevicizumab in HER2-low breast cancer with brain metastasis.

DETAILED DESCRIPTION:
This is a Phase II, open-label, multicenter, randomized controlled trial (THUMB study) comparing the efficacy and safety of trastuzumab deruxtecan (T-DXd) with or without bevacizumab for HER2-low expressing breast cancer with brain metastases. Patients receiving treatment in the metastatic setting must not have received more than 3 lines of therapy (HR-positive patients must have received a CDK4/6 inhibitor). Participants are randomized in a 1:1 ratio to receive treatment with T-DXd combined or not combined with bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG score of 0 to 1.
2. Expected survival period greater than 12 weeks.
3. Histologically confirmed invasive HER2-low expressing breast cancer (specific definition: breast cancer patients with low expression of human epidermal growth factor receptor 2 (HER-2) as determined by pathological testing. Specifically: HER2 IHC 1+ or HER2 IHC++ with FISH/CISH negative. All specimens must be verified by the pathology department of the research participating center.
4. Tumor stage: recurrent or metastatic breast cancer; local recurrence must be confirmed by the researcher to be unable to undergo radical surgical resection.
5. Patients must have at least one lesion that has not previously received radiation therapy (measurable and/or non-measurable).
6. MRI or CT shows brain metastasis and meets one of the following conditions:

   i) Untreated brain parenchymal metastasis found by imaging screening; ii) Previously locally treated stable or progressive brain parenchymal metastasis and meets one of the following conditions:a) Imaging stability ≥4 weeks; b) New brain parenchymal metastasis found by MR or CT.
7. Received no more than 2 lines of chemotherapy after metastasis.
8. HR-positive patients must have previously received CDK4/6 inhibitor treatment, whether in the adjuvant treatment phase or in the recurrent metastatic phase.
9. Never used T-DXd or bevacizumab before.
10. The main organ functions are basically normal, meeting the following conditions:
11. Blood routine examination standards must comply with: HB≥90g/L (not transfused within 14 days); ANC≥1.5×10^9/L; PLT≥75×10^9/L;
12. Biochemical examination must comply with the following standards: TBIL≤1.5×ULN (upper limit of normal); ALT and AST≤3×ULN; if there is liver metastasis, ALT and AST≤5×ULN; serum Cr ≤1.5×ULN, endogenous creatinine clearance rate ≥30mL/min.
13. Allowed to use mannitol, hormone therapy before enrollment, but the drug treatment dose can be stable for at least one week without the need for an increase.
14. Female subjects with reproductive capacity need to use one medically recognized contraceptive method during the study treatment period and for at least 3 months after the last use of the study drug.
15. Subjects voluntarily join this study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. Received more than 2 lines of chemotherapy.
2. Used T-DXd or bevacizumab.
3. Meningeal metastasis.
4. Brain metastasis requiring emergency intervention treatment, or brain metastasis requiring treatment with more than 3mg/d of dexamethasone or equivalent medication.
5. Clinical significant or uncontrolled cardiac disease history, including congestive heart failure, angina, myocardial infarction within the past 6 months, or ventricular arrhythmia.
6. Ongoing adverse reactions of grade >1 due to previous treatment. The exception is alopecia or those that the researcher believes should not be excluded. Such cases should be clearly documented in the investigator's notes.
7. Pregnant patients.
8. History of other malignancies within the past 5 years, excluding cured cervical carcinoma in situ, skin basal cell carcinoma, or skin squamous cell carcinoma.
9. Inability to swallow, chronic diarrhea, and intestinal obstruction, with multiple factors affecting drug intake and absorption.
10. Third space fluid accumulation (such as massive pleural effusion and ascites) that cannot be controlled by drainage or other methods.
11. Participated in another antitumor drug clinical trial within 4 weeks before the first administration of the study drug.
12. Long-term non-healing wounds or incompletely healed fractures.
13. Known HBV or HCV infection during the active phase or HBV DNA ≥500, or chronic phase with abnormal liver function.
14. Active primary immunodeficiency, known HIV test positive.
15. Uncontrolled infection requiring intravenous antibiotics, antiviral drugs, or antifungal drugs.
16. History of (non-infectious) ILD/pneumonia requiring steroids, currently having ILD/pneumonia, or unable to exclude suspected ILD/pneumonia on imaging during screening.
17. Pulmonary criteria:
18. Clinically significant pulmonary comorbidities, including but not limited to any underlying pulmonary disease (e.g., pulmonary embolism, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion, etc.) within 3 months of study recruitment.
19. Any autoimmune disease, connective tissue disease, or inflammatory disease (e.g., rheumatoid arthritis, Sjögren's syndrome, sarcoidosis, etc.) with recorded or suspected pulmonary involvement during screening. All detailed information about the disease should be recorded in the CRF for participants in the study.
20. Previous total pneumonectomy.
21. Allergic constitution, or known history of allergy to any component of the study regimen, or allergic to other monoclonal antibodies.
22. History of gastrointestinal bleeding within the past 6 months or a clear tendency for gastrointestinal bleeding, such as: esophageal varices at risk of bleeding, local active ulcer lesions, fecal occult blood ≥ (++) not eligible for enrollment; if fecal occult blood (+), gastroscopy is required;
23. Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days before participating in this study;
24. Urinalysis shows urine protein ≥++ or confirmed 24-hour urine protein quantitative >1.0g;
25. Hypertension, and blood pressure cannot be lowered to the normal range with antihypertensive drugs (systolic blood pressure >140mmHg, diastolic blood pressure >90mmHg).
26. Substance abuse or medical conditions that the researcher believes may interfere with the subject's participation in the clinical study or the assessment of the clinical study results.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) | 12 months
  Time to progressive disease (according to RECIST1.1)

SECONDARY OUTCOMES:
CNS Progression-free survival (CNS-PFS) | 12 months
  Time from enrollment to the first radiographic documented disease progression (PD) of all CNS target lesions (RANO-BM criteria) or death from any cause without progression was recorded.
Objective response rate (ORR) | 12 months
  Partial response is defined as a decrease by 30% or more in sums of longest diameter of measurable target lesions
CNS Objective response rate (CNS-ORR) | 12 months
  The proportion of patients with complete response (CR) and partial response (PR) evaluated as the best response observed from enrollment to progression of all CNS target lesions assessed according to RANO-BM criteria among the total number of patients who could be evaluated.
Overall survival (OS) | 12 months
  Time from the enrollment to death of any cause
Safety and Tolerability | 12 months
  Safety and Tolerability Will be Assessed According to Standard (CTCAE Version 5.0) Toxicity Reporting Criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided